CLINICAL TRIAL: NCT05397990
Title: Investigating the Impact of Exercise on Hippocampus-dependent Cognition and the Gut Microbiota in a Healthy, Middle-aged Population: The NeuroFit Study
Brief Title: The Impact of Exercise on Hippocampus-dependent Cognition and the Gut Microbiota
Acronym: NeuroFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Reta Lila Weston Trust (Unknown); University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HR/DP-21/22-28287
Record Dates: First submitted 2022-05-20; First posted 2022-05-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Decline
Keywords: Cognition; Pattern separation; Memory function; Gut microbiota; Exercise; Neurogenesis; Lifestyle
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 12 weeks exercise intervention. 3 times a week, 45 minutes per session, 30 minutes of exercise.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Continue with habitual routine. Take part in weekly online socials with others in the control group.

INTERVENTIONS:
Behavioral: Exercise — 12 weeks of moderate intensity exercise, three times a week.
  Arms: Exercise

SUMMARY:
The NeuroFit study will be investigating the impact of exercise on global cognition, hippocampus-dependent memory function and the gut microbiota in a middle-aged population.

DETAILED DESCRIPTION:
Main research question: Does exercise have an impact on global cognition, hippocampus-dependent memory function and the gut microbiota in a middle-aged human population?

Middle-age is a critical time for cognitive/mood changes and precedes prodromal dementia, which is mediated by changes in neuroplasticity and altered gut microbiota. This period of the lifespan is also associated with weight gain, decline in metabolism and physical fitness. Yet, it is unclear if cognitive and mood changes can be ameliorated in response to exercise and the role of gut microbiota.

The hippocampus plays a role in cognition and mood and is vulnerable to gut-mediated and metabolic changes. It is capable of generating new neurons from neural stem cells throughout life. This is a modifiable process of neuroplasticity called adult hippocampal neurogenesis (AHN), which decreases with age in the human and rodent brain. Exercise is a robust enhancer of AHN and attenuates deficits in the aged brain. Rodent studies have shown that AHN underlies antidepressant effects and certain forms of memory. In particular, pattern separation, the ability to discriminate between similar experiences or environments. A reduced ability to pattern separate is evident in older individuals and is an early symptom in mild cognitive impairment, which can present during middle-age. Moreover, pattern separation has been shown to be impaired and AHN decreased in middle-aged relates compared to young rats. Pattern separation has also been implicated as critically sensitive to exercise. However, the potential for exercise to prevent/reverse a deficit in AHN and pattern separation in middle-age has not yet been investigated. A major gap in knowledge is the identification of the mechanisms underlying cognitive impairment in middle-age, and how modulating factors, such as exercise, could attenuate them.

The investigators propose that the composition of the gut microbiota and their metabolites in middle-age may predict reduced AHN and pattern separation, which may be rescued/improved by exercise, and is thus a key mechanistic target for investigation. In support, ageing is associated with a decline in gastrointestinal function and a change in microbiota composition. Middle-age is particularly vulnerable for gut microbiota compositional and metabolite changes coupled with neuroinflammation in mice, and that these effects are modified in response to prebiotic supplementation. An altered gut microbiota is associated with low mood/depressive behaviour through metabolic changes, and germ-free mice display an aberrant increase of neurogenesis. Moreover, preliminary data show that gut microbiota depletion (induced by long-term antibiotic administration) leads to a decrease in pattern separation and AHN, albeit in young adult rats.

Accumulating evidence suggests that exercise can change gut microbial composition and serum metabolites. Interestingly, human and rats present the same metabolic signature in plasma after exercise. Moreover, the effects of exercise on metabolic profiles are transmissible via faecal microbiota transplantation (FMT). Considering the gut microbiota (i) is sensitive to exercise and age, (ii) regulates AHN and, (iii) is involved in pattern separation and mood, the investigators propose that the gut microbiome-AHN communication is important in maintaining hippocampal integrity and cognitive function during middle-age.

Aim The overall aim of the NeuroFit study is to develop and test the impact of a group-based exercise intervention to identify specific gut microbiota and metabolic signatures that may influence cognitive and mood changes in middle-aged adults.

Hypothesis Reduced pattern separation in middle age can be rescued/improved by exercise accompanied by changes in the gut microbiota and related metabolites.

Objectives The NeuroFit study has 3 main objectives.

1. Determine the impact of a 12-week exercise intervention (30 minutes, 3 days a week) compared to a control group (continued habitual behaviour) in healthy, middle-aged participants on cognition and mood.
2. Identify specific gut microbiota and metabolic signatures in middle age which is responsive to exercise and predictive of cognitive and mood changes in a randomised controlled trial.
3. Assess the impact of exercise on neuropsychiatric symptoms, serum BDNF, dietary intake, quality of life, habitual physical activity, cardio-respiratory fitness, anthropometry and cardiometabolic health on cognition and mood.

ELIGIBILITY:
Inclusion Criteria:

1. 45 - 65 years of age.
2. BMI 20 - 30.
3. Does less than 90 minutes of moderate to vigorous physical activity per week and does not have a regular exercise routine(captured by self-reported measures)

Exclusion Criteria:

1. Subject is unable to understand the participant information sheet.
2. Subject is unable to provide written informed consent.
3. Subject is unable to understand and/or completely perform the cognitive testing.
4. Impaired vision that is not corrected.
5. Subject is a smoker.
6. Does not agree to maintain their habitual dietary routine.
7. Unwilling to provide blood and stool samples.
8. Is not in general good health on the basis of medical history.
9. Unable to engage in a structured exercise program as determined by the physical activity readiness questionnaire (PARQ).
10. Unwilling to engage in the prescribed exercise program 3 times a week.
11. Subject is pregnant, lactating or planning pregnancy.
12. Recent history (previous 2 years) or currently diagnosed with a significant psychiatric disorder including major depressive disorder, anxiety, bipolar disorder, schizophrenia or any other Diagnostic Statistical Manual (DSM)-IV Axis I disorder.
13. Subject has significant acute or chronic co-existing cardiovascular, respiratory, gastrointestinal illness or liver disease.
14. Subject has had major GI surgery including bariatric surgery (excluding appendectomy and cholecystectomy).
15. History of cancer in the last 5 years (excluding melanoma).
16. Subject has significantly out of range blood test results from screening visit.
17. History of or currently diagnosed with a functional GI disorder including inflammatory bowel disease (including Crohn's disease and ulcerative colitis), coeliac disease, lactose intolerance and clinical diagnosis of irritable bowel syndrome.
18. Subject has irritable bowel syndrome, functional diarrhoea or functional constipation as determined by the Rome IV.
19. Subject has any neurological disorder that could produce cognitive deterioration including Alzheimer's disease, Parkinson's disease, and stroke.
20. Subject has a neurodevelopmental disorder that impacts ability to take part in cognitive testing and/or memory function.
21. History of traumatic brain injury, stroke or any other medical conditions causing cognitive impairment.
22. Subject has uncontrolled epilepsy or is prone to fainting.
23. Subject has an eating disorder.
24. History of or currently diagnosed with a metabolic disorder including type 1 and type 2 diabetes mellitus.
25. Subject is unwilling to stop taking prebiotics or probiotics for at least 4 weeks prior to commencing the study.
26. Known or suspected of alcohol abuse defined as > 14 drinks per week (1 drink = 1 pint of beer, 1 large glass of wine or 50 ml spirit).
27. Subject has a sleep disorder or an occupation where sleep during the overnight hours is irregular.
28. Subjects routinely taking psychoactive medications, laxatives, enemas, antibiotics, anticoagulants, NSAIDs, proton pump inhibitors and unwilling to stop at least 4 weeks prior to commencing the study.
29. Subjects taking the following prescription medications: Statins, Metformin, Donepezil (Aricept), Galantamine (Reminyl), Rivastigmine (Exelon), Tacrine (Cognex), Memantine (Namenda), Selegiline (Eldepryl) or any other medication for cognitive impairment.
30. Subject has a condition the chief investigator believes would interfere with their ability to provide informed consent, comply with the study protocol, may confound the interpretation of study results, or put the subject at undue risk.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Mnemonic Similarity Task | Change from baseline pattern separation and recognition memory at 12 weeks
  Pattern separation and recognition memory
Mnemonic Similarity Task | Change from baseline pattern separation and recognition memory at 24 weeks
  Pattern separation and recognition memory

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 | Change from baseline mood at 12 weeks
  Mood score Scoring scale: 0 - 27 Lower scores = better outcome.
Patient Health Questionnaire 9 | Change from baseline mood at 24 weeks
  Mood score Scoring scale: 0 - 27 Lower scores = better outcome.
Gut microbiome composition | Change from baseline composition at 12 weeks
  Taken from participant stool samples. Measured using shotgun metagenomic sequencing.
Metabolomic profile - Serum | Change from baseline profile at 12 weeks
  Metabolomic screen of participant serum samples at MS-Omics (Denmark)
Metabolomic profile - Gut microbiota | Change from baseline profile at 12 weeks
  Metabolomic screen of participant stool samples at MS-Omics (Denmark)
Short Form 12 | Change from baseline quality of life at 12 weeks
  Quality of life scale Scoring scale: 0 - 100 Higher scores = better outcome.
Short Form 12 | Change from baseline quality of life at 24 weeks
  Quality of life scale Scoring scale: 0 - 100 Higher scores = better outcome.
Cardiorespiratory fitness | Change from baseline fitness at 12 weeks
  3 minute step test
Cardiorespiratory fitness | Change from baseline fitness at 24 weeks
  3 minute step test
Bone derived neurotrophic factor (BDNF) | Change from baseline BDNF levels at 12 weeks
  Measured from participant serum sample using an enzyme-link immunoabsorbant assay
Bone derived neurotrophic factor (BDNF) | Change from baseline BDNF levels at 24 weeks
  Measured from participant serum sample using an enzyme-link immunoabsorbant assay
Nutritional intake | Change from baseline nutritional intake at 12 weeks
  4 day food diary
Nutritional intake | Change from baseline nutritional intake at 24 weeks
  4 day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Thuret, PhD, Principal Investigator — King's College London; Brendon Stubbs, PhD, Principal Investigator — King's College London
Locations (1):
- Curie Kim, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code